CLINICAL TRIAL: NCT01788293
Title: Fluid Management Based on Pleth Variability Index (PVI) Monitoring During High-risk Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Problem with recruiting
Sponsor: Hospital Regional de Presidente Prudente (Other)
Responsible Party: Principal Investigator, Edmundo Pereira de Souza Neto, Professeur, MD, Hospital Regional de Presidente Prudente
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PVI - HR
Record Dates: First submitted 2013-02-06; First posted 2013-02-11 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Fluid Loss
Keywords: Fluid management; Pleth Variability Index (PVI); monitoring; high-risk surgery

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Active Comparator): Intervention group will receive hydroxyethylstarch 6% bolus in order to minimize and maintain PVI below 14 %.
  Interventions: Other: Intervention group
- Control group (No Intervention): Control group will receive fluid at the discretion of the anesthetist

INTERVENTIONS:
Other: Intervention group — Control group will receive per-operative fluid at the discretion of the anesthetist, whereas Intervention group will receive additional hydroxyethylstarch 6% (HES) bolus in order to minimize and maintain PVI below 14 %.
  This PVI cut-off value was chosen according to previous reports [Cannesson et al., 2008; Zimmermann et al., 2010].
  During the postoperative period, both groups were managed by intensivists (in the ICU) and clinicians (in the wards) not involved in the intraoperative management or in data collection. These individuals were not informed of patient allocation.
  Arms: Intervention group

SUMMARY:
Oximetry monitoring is common practice in patients undergoing anesthesia. PVI continuous evaluation may be a possibility of agility and ease of obtaining accurate information about the state of cardiovascular responsiveness to volume expansion.

This prospective and randomized study will try to demonstrate that the assessment of PVI is a simple and cost-saving method as compared to cardiac output or oxygen delivery monitoring technologies. Such a simple approach has therefore the potential for widespread application as it is not routinely feasible for anesthetists to use cardiac output or oxygen delivery monitoring technologies in many institutions, as well as in many countries.

DETAILED DESCRIPTION:
Introduction

Several studies have shown that cardiac output optimization improve postoperative outcome and to decrease the cost of surgery [Boyd et al., 1993; Gan et al., 2002; Kern & Shoemaker, 2002 ; Pearse et al., 2005 ; Poeze et al., 2005 ; Sinclair et al., 1997; Wakeling et al., 2005].

Respiratory variations in the arterial pulse pressure and in the pulse oximetry plethysmographic waveform amplitude have been extensively studied in mechanically ventilated patients, and have been demonstrated to be sensitive to changes in ventricular preload as well as reliable predictors of fluid responsiveness in adults [Cannesson et al 2007; Cannesson et al., 2008; Natalini et al., 2006; Solus-Biguenet et al., 2006; Zimmermann et al., 2010].

A few studies have evaluated the impact of a pulse-pressure-variations-guided fluid management on perioperative outcome [Buettner et al., 2008; Fukui et al., 2007; Fukui et al., 2009; Kobayashi et al., 2008; Lopes et al., 2007; Mayer et al, 2009; Oubaha & Poelaert, 2009; Sakamoto et al., 2009]. However, results from these studies are not conclusive and further studies are required to better explore this topic [Cannesson, 2010].

Pulse oximeters are part of the routine monitoring during anesthesia and in the intensive care unit [Dorlas & Nijboer, 1985]. The main interest of the pulse oxymeter is to display arterial oxygenation continuously. Pleth variability index (PVI) is an automatic measure of the dynamic change in perfusion index (PI) that occurs during a complete respiratory cycle. PVI is provided currently by one pulse oximeter manufacturer (Masimo Radical 7 ™, Masimo Corporation, Irvine, CA, USA). The PVI calculation measures changes in PI over a time interval sufficient to include one or more complete respiratory cycles as and is displayed continuously [Cannesson et al., 2008; Zimmermann et al., 2010]. PVI quantifies the variability in plethysmograph waveform due to respiration and is thought to be a surrogate measure of intravascular volume [Cannesson et al., 2008; Zimmermann et al., 2010]. Cannesson et al. reported that a PVI value above 14% predicted fluid responsiveness [Cannesson et al., 2008]. Therefore, the clinical and intra-operative goal of "maximizing stroke volume by volume loading" can be achieved by reducing PVI below 14 % [Cannesson et al., 2008; Zimmermann et al., 2010]. Forget et al [2010] demonstrated that PVI based goal-directed fluid management reduced the volume of intraoperative fluid infused and reduced intraoperative and postoperative lactate levels. However, to our knowledge there is no study that evaluate the impact of PVI guided fluid management on perioperative outcome.

Materials and Methods

Patients This procol has been approved by the local Ethics Committee (Hospital Regional de Presidente Prudente Presidente Prudente, São Paulo, Brazil). The written informed consent will be obtained from each patient. Adults patients underwent high-risk surgery will be selected and randomized to either a control group (group C) or an intervention group (group I).

Patients will be selected according to a pre-operative decision (by the surgeon and the intensivist) that post-operative care would be undertaken in the ICU because of co-morbidities or/and the surgical procedure. Patients < 18 years, with cardiac arrhythmias, with a body mass index > 40, and those undergoing surgery with an open thorax, neurosurgery or emergency surgery, will be excluded.

Intraoperative monitoring

On the day of surgery, they will receive their respective medication in association with anesthetic premedication. Immediately after the arrival in the operating room heart rate, pulse oximetry, blood pressure and capnography will be monitored with a multiparameter bedside monitor (DX 2023, Dixtal™, São Paulo, Brazil). A 20-G catheter line (Smith Medical International™, Lancashire, Uk) will be inserted in the radial artery for continuous arterial pressure measurement and recording. The radial catheter will be connected to a Dixtal® DX 2023 monitor (São Paulo, Brazil).

The patients will be anesthetized with loading doses of propofol (2 mg/kg), sufentanil (0,2 - 0,3 µg/kg) and atracurium (0.6 mg/kg). Anesthesia will be maintained by infusion of the same products. After induction of anesthesia, patients underwent tracheal intubation. Artificial ventilation will be provided by a Fabius plus ™ ventilator (Dräger™, Lübeck, Germany) (respiration rate = 12 strokes/min, tidal volume = 8 to 10 ml/kg).

Each respiratory cycle will be identified from the capnogram, systolic and diastolic arterial pressures will be measured on a beat-to-beat basis. In patients of intervention group PVI values will be determined over each respiratory cycle (Masimo Radical 7 ™, Masimo Corporation, Irvine, CA, USA).

Protocol Randomization will be done pre-operatively using sealed envelopes. During the surgical procedure, patients will be managed according to our institution's standard of care. Group C will receive per-operative fluid at the discretion of the anesthetist, whereas group I will receive additional hydroxyethylstarch 6% (HES) bolus in order to minimize and maintain PVI below 14 %. This PVI cut-off value was chosen according to previous reports [Cannesson et al., 2008; Zimmermann et al., 2010].

During the postoperative period, both groups were managed by intensivists (in the ICU) and clinicians (in the wards) not involved in the intraoperative management or in data collection. These individuals were not informed of patient allocation.

Data collection

Over the study period all data will be collected prospectively and patients will be followed up until hospital discharge. Pre and intraoperative data collection will be undertaken by one of the investigators, whereas post-operative data collection will be undertaken by another, who was not aware of the allocation group. Before surgery, sex, age, weight, height, history of renal failure requiring dialysis or not, cirrhosis, chronic obstructive pulmonary disease, hypertension, peripheral vascular disease, coronary artery disease, other cardiac disease, diabetes mellitus, and cerebrovascular disease will be recorded. The body mass index will be calculated according to the standard formula (BMI = weight/height2). Serum creatinine, prothrombin time, hemoglobin, and platelets will be obtained from routine pre-operative biological tests. During the surgical procedure, tidal volume, ventilatory frequency, infused volume of crystalloid solutions, HES, and blood products will be recorded. Heart rate, mean arterial pressure, percutaneous arterial oxygen saturation, and hemoglobin will be collected both at the beginning and the end of the surgical procedure. The duration of surgery will be also recorded. After the surgical procedure, the following parameters will be collected both at ICU admission and 24h later: mean arterial pressure, heart rate, percutaneous arterial oxygen saturation. During the 24h following ICU admission, venous lactate will be measured every 6h and the mean lactate value will be calculated over the first 24h ICU period. The need for continuous vasoactive (dobutamine or/and norepinephrine) support will be recorded.

Postoperative ICU infections (pneumonia, abdominal, urinary tract, line related sepsis and wound infections), respiratory complications (pulmonary embolism, acute lung injury, and respiratory support > 24h exclusive of acute lung injury), cardiovascular complications (arrhythmia, hypotension, acute pulmonary edema, acute myocardial infarction, stroke, and cardiac arrest exclusive of fatal outcome), abdominal complications (clostridium difficile diarrhoea, acute bowel obstruction, upper gastro-intestinal bleed, and anastomotic leak), hematologic complications (platelet count < 100000/µl or prothrombin time > 1.5 times control), and renal complications (urine output < 500 ml/day or serum creatinine > 170 µmol/L or dialysis for acute renal failure) were collected according to criteria previously used by other investigators [Bennett-Guerrero et al., 1999; Gan et al., 2002; Lopes et al., 2007; Pearse et al., 2005].

Statistical analysis

Data will be analyzed comparing patients in group C with those in group I on an intention-to treat basis. The primary outcome measure will be the duration of postoperative hospital stay. On the basis of our own hospital registry, the mean duration of postoperative hospital stay in group C is a priori estimated at 15 ± 7 days (median ± median absolute deviation). According to previous publications we postulated that the mean duration of postoperative hospital stay in group I could be 35% lower [Lopes et al., 2007; Mythen & Webb, 1995; Sinclair et al., 1997]. A sample size of 35 patients in each group was calculated for a 0.05 difference (two sided) with a power of 80% [Schulz & Grimes, 2005]. An intermediate analysis after the enrolment of the first 35 patients was planed, in order to readjust the population sample size if necessary. Secondary outcome measures were the number of post-operative complications per patient, as well as the duration of mechanical ventilation and ICU stay. Results are expressed as median ± median absolute deviation. The median absolute deviation is a variation of the average absolute deviation that is even less affected by outlying values because these values have less influence on the calculation of the median than they do on the mean. In general, for data with extreme values, the median absolute deviation or interquartile range can provide a more stable estimate or variability than the standard deviation.

The Mann-Whitney U test was used to compare between groups patient characteristics as well as the duration of mechanical ventilation, ICU stay and hospital stay. In group I, the effects of volume expansion with HES administration in PVI will be assessed using a nonparametric Wilcoxon rank sum test within each group of patients. A Fisher exact test was performed to compare nominal data. Linear correlations were tested using the Spearman rank method. A p-value lower than a 0.05 chosen level is regarded as statistically significant. All statistical analyses are performed using the StatView TM software for Windows (version 4.57, Abacus Concepts Inc., Berkeley, CA, USA).

ELIGIBILITY:
Inclusion Criteria:

* Adults patients underwent high-risk surgery
* obtained the written informed consent
* patients under general anesthesia and mechanical ventilation

Exclusion Criteria:

* Patients with cardiac arrhythmias
* Patients < 18 years
* Patients with a body mass index > 40
* Patients undergoing surgery with an open thorax, neurosurgery or emergency surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-02; Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the duration of postoperative hospital stay. | An intermediate analysis after the enrolment of the first 35 patients was planed, in order to readjust the population sample size if necessary.
  On the basis of our own hospital registry, the mean duration of postoperative hospital stay is a priori estimated at 15 ± 7 days (median ± median absolute deviation).

SECONDARY OUTCOMES:
Secondary outcome measures were the number of post-operative complications per patient | 30 days (plus or minus 5 days)

CONTACTS AND LOCATIONS:
Overall Officials: Edmundo P Souza Neto, PhD, MD, Principal Investigator — Hospital Regional de Presidente Prudente
Locations (1):
- Hospital Regional de Presidente Prudente, Presidente Prudente, São Paulo, Brazil